CLINICAL TRIAL: NCT03268213
Title: Fecal Microbial Transplantation in Patients With Medication Refractory Clostridium Difficile and/or Ulcerative Colitis or Indeterminate Colitis
Brief Title: Fecal Microbial Transplantation for C. Difficile and/or Ulcerative Colitis or Indeterminate Colitis
Acronym: FMT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Anupama Chawla, Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 479696
Record Dates: First submitted 2016-03-22; First posted 2017-08-31 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Clostridium Difficile Infection; Ulcerative Colitis; Indeterminate Colitis
MeSH Terms: conditions — Clostridium Infections; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: FMT is offered as a treatment to eligible patients
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal microbial transplantation (Experimental): Treated with fecal microbial transplantation
  Interventions: Biological: Fecal Microbial Transplantation

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — Fecal microbial transplant is offered as treatment option to eligible patients. Donors selected by the patients will be screened by questionnaire and by blood and stool tests for potential transmissible pathogens.
  The stool filtrate will be administered in the ileum and/or cecum via colonoscopy
  Other Names: FMT

SUMMARY:
Fecal Microbiota Transplantation will be offered to eligible C. difficile patients (does not require Investigational New Drug designation) and to eligible ulcerative colitis or indeterminate colitis patients as Investigational New Drug treatment

DETAILED DESCRIPTION:
The following hypothesis will be tested in this study:

1. Fecal microbiota transplantation is a safe, tolerable, and efficacious procedure for C. difficile patients and is a safe and tolerable procedure for ulcerative colitis and indeterminate colitis patients.
2. The fecal microbial diversity, composition and function in stool recipients after fecal transplantation will change to a similar microbial diversity, composition and functionality as found in donor stool.

Primary objectives:

1. To determine the short term safety and tolerability of fecal microbiota transplantation in patients with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis up to 12 weeks post-transplant.

Secondary objectives:

1a. To determine the long term safety and tolerability of fecal microbiota transplantation up to 1 year post-transplant in patients with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

1b. To determine the efficacy of fecal microbiota transplantation in patients with recurrent or refractory Clostridium difficile defined as no recurrence of C. difficile within one year.

2. To compare microbial diversity in healthy donor stools compared to pre-FMT recipient stools collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

3. To compare microbial composition in healthy donor stools compared to pre-FMT recipient stools from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

4. To compare microbial function in healthy donor stools compared to pre-FMT recipient stools from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

5. To compare microbial diversity in healthy donor stools and pre-FMT recipient stools with 1 week post-transplant recipient stool samples collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

6. To compare microbial composition in healthy donor stools and pre-FMT recipient stools with 1 week post-transplant recipient stool samples collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

7. To compare microbial function in healthy donor stools and pre-FMT recipient stools with 1 week post-transplant recipient stool samples collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

8. To compare microbial diversity in healthy donor stools and pre-FMT recipient stools with 12 week post transplant recipient stool samples collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

9. To compare microbial composition in healthy donor stools and pre-FMT recipient stools with 12 week post transplant recipient stool samples collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

10. To compare microbial function in healthy donor stools and pre-FMT recipient stools with 12 week post transplant recipient stool samples collected from patients (recipients) with recurrent or refractory Clostridium difficile and medication refractory Ulcerative colitis or indeterminate colitis.

11. Stool calprotectin levels will be measured in the recipient at baseline pre-FMT, 1 week and 12 weeks post FMT to determine if FMT causes a statistically significant change.

ELIGIBILITY:
For C. difficile patients/recipients only:

Inclusion:

1. Patient is 7 years of age or older. 2. One of the following: 2a. At least two recurrences (total three CDI infections) of mild to moderate C. difficile (<6 diarrheal stools/day) diagnosed by positive toxin PCR or EIA after completing standard medical therapy with metronidazole, vancomycin or fidaxomicin.

2b. At least two episodes of severe C. difficile infection (>6 diarrheal stools/day requiring hospitalization and associated with significant morbidity).

2c. Moderate C. difficile infection (3-6 diarrheal stools/day not responding to successive standard therapy, e.g. metronidazole, vancomycin and/or fidaxomicin) lasting at least 28 days.

2d. Severe and/or fulminant C. difficile colitis (> 6 diarrheal stools/day) with no response to standard therapy after 48 hours.

Exclusion:

1. younger than 7 year old
2. scheduled for abdominal surgery within the next 12 weeks
3. had major abdominal surgery within the past 3 months
4. pregnancy
5. Hemoglobin < 6 g/dL
6. absolute neutrophil count less than 1500/mm3
7. known diagnosis of graft vs. host disease
8. used an investigational drug within the past 2 months
9. used a TNFα agonist within the past 2 weeks
10. diagnosed with Bacteremia within the past 4 weeks

For patients with ulcerative and indeterminate colitis only:

Inclusion:

1. Patient is 7 years of age or older.
2. One of the following:

2a. treated with steroid therapy for at least one month. 2b. treated with immunomodulatory therapy for at least one month 2c. treated with biological therapy for at least one month.

Exclusion:

1. younger than 7 years old
2. scheduled for abdominal surgery within the next 12 weeks
3. had major abdominal surgery within the past 3 months
4. pregnancy
5. Hemoglobin < 6 g/dL
6. absolute neutrophil count less than 1500/mm3
7. known diagnosis of graft vs. host disease
8. used an investigational drug within the past 2 months
9. used a TNFα agonist within the past 2 weeks
10. diagnosed with Bacteremia within the past 4 weeks
11. previous FMT

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 9 years
  Number of participants with treatment-related adverse events with grade greater than 2 within one year after FMT will be reported.
  Safety will be assessed as a report of no new medical condition after the transplant, Tolerability, as recorded by report of no serious adverse events after the transplant and Efficacy of the procedure will be recorded as improvement in clinical symptoms during any clinically indicated colonoscopies after the transplant as compared to before transplant
  C. Diff patients will have a negative C. diff test report after the transplant as an out come measure.

SECONDARY OUTCOMES:
To measure the effect of fecal microbial transplantation on microbial diversity in healthy donor stools compared to pre-FMT, 1 week post FMT, and 12 weeks post-FMT recipient stools. | 10 years
  Fecal DNA samples will undergo V3-V4 16S rRNA sequencing. Operational taxonomic units (OTUs) will be produced by clustering sequences with identical taxonomic assignments. Alpha diversity indices (e.g. Chao1, Shannon complexity H, Shannon Evenness H/Hmax) will be calculated inferred through 1000 replicate resamplings using Explicet. Beta diversity (Bray-Curtis and Jaccard distances) will be calculated for the recipient Pre-FMT, 1 week post-FMT and 12 weeks post-FMT as compared to their pared donor using the adonis function in the R vegan package at the phyla, family and genus level. A linear mixed model will be used to compare alpha-diversity (ShannonH) and beta-diversity (Bray-Curtis and Jaccard distance) between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
To measure the effect of fecal microbial transplantation on microbial composition in healthy donor stools compared to pre-FMT, 1 week post FMT, and 12 weeks post-FMT recipient stools. | 10 years
  Fecal DNA samples will undergo V3-V4 16S rRNA sequencing. Operational taxonomic units (OTUs) will be produced by clustering sequences with identical taxonomic assignments. Linear mixed models analyses on individual OTUs at the genus level will be conducted on 105 OTUs after eliminating OTUs with an average relative abundance of < 0.001% in the donor and recipient pre-FMT samples, and after discarding OTUs where more than 75% of the samples had a zero count. To compare the relative abundance of each OTU between timepoints before and after FMT [pre-transplant recipient, 1-wk. post-FMT recipient, 3-mos. post-FMT recipient] and each disease group, a generalized linear mixed model (GLMM) or generalized estimating equation (GEE) will be used by taking the actual counts of each OTU as the outcomes that were assumed to follow a negative binomial distribution. The p-values will be adjusted for multiple comparisons by the Bonferroni correction or by the Benjamin-Hochberg method (FDR < 0.05).
To measure the effect of fecal microbial transplantation on microbial function using shotgun DNA metagenomic in healthy donor stools compared to pre-FMT, 1 week post FMT, and 12 weeks post-FMT recipient stools. | 10 years
  Fecal DNA samples will undergo shotgun DNA metagenomics sequencing. After removing human sequences, the Reads per kilobase gene length (RKP) will be calculated using HUMANN2 software for individual bacterial proteins/enzymes and pathways. . A linear mixed model will be used to compare RPK associated with pathways and individual proteins between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.Linear mixed models analyses on the RPK associated with individual genes and pathways will be analyzed using linear mixed models between timepoints before and after FMT [pre-transplant recipient, 1-wk. post-FMT recipient, 3-mos. post-FMT recipient] and each disease group, a generalized linear mixed model (GLMM) or generalized estimating equation (GEE) were used by taking the actual RPK as the outcomes that will be assumed to follow a negative binomial distribution.
To measure the effect of fecal microbial transplantation on microbial function using bacterial metatranscriptomic sequencing | 10 years
  Fecal RNA samples will undergo bacterial metatranscriptomic RNA sequencing. After removing human sequences, the Reads per kilobase transcript (RKP) will be calculated for individual bacterial proteins/enzymes and pathways. A linear mixed model will be used to compare RPK associated with pathways and individual proteins between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
To measure the effect of fecal microbial transplantation on microbial function using targeted metabolomic assays. | 10 years
  Fecal samples will undergo extraction for targeted metabolomics analysis of short chain fatty acids (micrograms/gram stool) using gas chromatography-mass spectrometry, and of bile acids (microgram/gram stool) using liquid chromatography-mass spectrometry. A linear mixed model will be used to compare respectively short chain fatty acid and bile acid metabolites between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
Determine if FMT causes a statistically significant change in recipient fecal calprotectin levels | 10 years
  Fecal calprotectin (microgram/gram stool) levels will be measured as in the recipient at baseline pre-FMT, 1 week, and 12 weeks post FMT. A linear mixed model will be used to compare fecal calprotectin levels between each timepoint (FMT) and each disease group (Group). P-values less than 0.05 were considered as statistically significant.
Determine number of C. difficile recipients who have recurrent C. difficile within a year after fecal microbial transplant | 10 years
  Currently the efficacy of colonoscopic FMT is approximately 90% after 12 weeks. However it may be lower with patients who also have inflammatory bowel disease. We will quantify the efficacy of fecal microbial transplant on C. difficile recurrence within a year in patients with C. difficile without inflammatory bowel diseases, C. difficile with Crohn's disease and C. difficile with ulcerative or indeterminate colitis.

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Chawla, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mintz M, Khair S, Grewal S, LaComb JF, Park J, Channer B, Rajapakse R, Bucobo JC, Buscaglia JM, Monzur F, Chawla A, Yang J, Robertson CE, Frank DN, Li E. Longitudinal microbiome analysis of single donor fecal microbiota transplantation in patients with recurrent Clostridium difficile infection and/or ulcerative colitis. PLoS One. 2018 Jan 31;13(1):e0190997. doi: 10.1371/journal.pone.0190997. eCollection 2018. PMID 29385143

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT03268213/Prot_ICF_002.pdf